CLINICAL TRIAL: NCT01085071
Title: GRIP-COMPASS Trial: Computer-driven Glucose and Potassium Regulation Program in Intensive Care Patients With COMparison of PotASSium Targets Within normokAlemic Range
Brief Title: Comparison of Two Potassium Targets Within the Normal Range in Intensive Care Patients
Acronym: GRIP-COMPASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Miriam Hoekstra, MD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRIP-COMPASS trial
Record Dates: First submitted 2010-03-01; First posted 2010-03-11 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Thoracic Surgery; Cardiac Surgery; Critically Ill
Keywords: intensive care unit; potassium; atrial fibrillation; cardiac surgery; Critically ill patients post CABG and/or valvular surgery; Critically ill patients not post CABG and/or valvular surgery; coronary artery bypass graft
MeSH Terms: conditions — Critical Illness; Atrial Fibrillation | interventions — Potassium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal-high potassium (NHP) (Active Comparator): A potassium target of 4.5 mmol/L.
  Interventions: Drug: Potassium Chloride
- Normal-low potassium (NLP) (Active Comparator): A potassium target of 4.0 mmol/L.
  Interventions: Drug: Potassium Chloride

INTERVENTIONS:
Drug: Potassium Chloride — KCl is continuously administered and titrated towards a Normal-high Potassium (4.5 mmol/L)
  Arms: Normal-high potassium (NHP)
Drug: Potassium Chloride — KCl is continuously administered and titrated towards a Normal-low Potassium (4.0 mmol/L)
  Arms: Normal-low potassium (NLP)

SUMMARY:
Rationale: It is well known that distinctly abnormal blood potassium values can cause serious complications such as cardiac arrhythmias. Although potassium regulation is generally considered important, hardly any research has been done about potassium regulation in intensive care patients. The investigators hypothesize that different potassium target-values, within the as normal accepted range, may have different effects in critically ill patients.

Study design: A prospective trial comparing two different potassium target-values. Potassium will be tightly regulated with the already fully operational GRIP-II computer program.

Study population: 1200 adult patients admitted at the thoracic intensive care unit of the University Medical Center Groningen.

Intervention: Comparison between two variations of standard therapy: potassium target-value of 4.0 mmol/L versus 4.5 mmol/L.

Main study parameters/endpoints: The primary endpoint is the incidence of atrial fibrillation or atrial flutter from ICU-admission to hospital discharge. Secondary endpoints are serum levels of potassium and the other main electrolytes, renal function and renal potassium excretion, the relation with insulin and glucose, the cumulative fluid balance, (ICU) length of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the thoracic and surgical ICU of the University Medical Center Groningen.
* Computerized potassium regulation with GRIP-II

Exclusion Criteria:

* Patients who are not potassium regulated with GRIP-II (patients who take their own meals).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
AFib or AFl in patients who underwent CABG (coronary artery bypass grafting) or valvular surgery. | First 7d after Intensive Care Unit admission or hospital discharge, whichever is earlier.
  Post-surgery AFib and AFl typically occur within days after surgery. AFib and AFl can only be reliably assessed during ICU stay and hospital stay. Therefore this outcome measure is not determined after hospital discharge.

SECONDARY OUTCOMES:
Potassium regulation within 3.5 to 5.0 mmol/L. | From Intensive Care Unit admission to hospital discharge.
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
AFib or AFl in other patients, i.e. patients who did not undergo CABG or valvular surgery. | First 7d after ICU-admission or hospital discharge, whichever is earlier.
  Post-surgery AFib and AFl typically occur within days after surgery. AFib and AFl can only be reliably assessed during ICU stay and hospital stay. Therefore this outcome measure is not determined after hospital discharge.
Biochemical disturbances including electrolytes (Na, K, Mg, Ca), blood gas analysis, lactate, renal function (creatinine, urea). | From ICU-admission to hospital discharge.
Cumulative fluid balance. | During ICU-stay.
Mortality and (ICU) length of stay. | ICU-mortality and hospital-mortality as well as 90-day mortality.
Glucose regulation | During ICU-admission.
  The relation with glucose levels and insulin administration

CONTACTS AND LOCATIONS:
Overall Officials: Felix Zijlstra, MD/PhD, Study Director — University Medical Center Groningen; Maarten WN Nijsten, MD/PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, University of Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Vogelzang M, Zijlstra F, Nijsten MW. Design and implementation of GRIP: a computerized glucose control system at a surgical intensive care unit. BMC Med Inform Decis Mak. 2005 Dec 19;5:38. doi: 10.1186/1472-6947-5-38. PMID 16359559
- [Background] Vogelzang M, Loef BG, Regtien JG, van der Horst IC, van Assen H, Zijlstra F, Nijsten MW. Computer-assisted glucose control in critically ill patients. Intensive Care Med. 2008 Aug;34(8):1421-7. doi: 10.1007/s00134-008-1091-y. Epub 2008 Apr 4. PMID 18389221
- [Background] Hoekstra M, Vogelzang M, Verbitskiy E, Nijsten MW. Health technology assessment review: Computerized glucose regulation in the intensive care unit--how to create artificial control. Crit Care. 2009;13(5):223. doi: 10.1186/cc8023. Epub 2009 Oct 16. PMID 19849827
- [Background] Hoekstra M, Vogelzang M, Drost JT, Janse M, Loef BG, van der Horst IC, Zijlstra F, Nijsten MW. Implementation and evaluation of a nurse-centered computerized potassium regulation protocol in the intensive care unit--a before and after analysis. BMC Med Inform Decis Mak. 2010 Jan 25;10:5. doi: 10.1186/1472-6947-10-5. PMID 20100342
- [Derived] Hoekstra M, Hessels L, Rienstra M, Yeh L, Lansink AO, Vogelzang M, van der Horst IC, van der Maaten JM, Mariani MA, de Smet AM, Struys MM, Zijlstra F, Nijsten MW. Computer-guided normal-low versus normal-high potassium control after cardiac surgery: No impact on atrial fibrillation or atrial flutter. Am Heart J. 2016 Feb;172:45-52. doi: 10.1016/j.ahj.2015.10.020. Epub 2015 Nov 11. PMID 26856215
- [Derived] Hoekstra M, Vogelzang M, van der Horst IC, Lansink AO, van der Maaten JM, Ismael F, Zijlstra F, Nijsten MW. Trial design: Computer guided normal-low versus normal-high potassium control in critically ill patients: Rationale of the GRIP-COMPASS study. BMC Anesthesiol. 2010 Dec 31;10:23. doi: 10.1186/1471-2253-10-23. PMID 21194419